CLINICAL TRIAL: NCT01600560
Title: Facilitating the Completion of the 3-Dose Series of HPV Vaccination in Males and Females
Brief Title: Facilitating Completion of HPV Vaccination
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 11-1551
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Adolescent Immunizations Among Clinic Population

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Social media

SUMMARY:
With the surge in use of electronic media among adolescents, a strategy that has been utilized to increase HPV4 uptake in girls has been reminder text messaging to their parents. To date, no published study has looked at the effectiveness of texting adolescents themselves (especially boys) rather than their parents OR compared texting to social network sites to increase HPV knowledge and uptake of HPV vaccination in boys. Interactive technology-based interventions targeted at youth are feasible in North Carolina for the following reasons: (1) through the NC Minors' Consent Law adolescents can consent to the prevention, diagnosis, and treatment of sexually transmitted diseases (N.C. Gen. Stat. § 90-21.5(a); and (2) many school based health centers can provide immunizations. Since HPV infection is a sexually transmitted infection, NC teens do not have to get consent for HPV prevention (i.e., vaccination).

To optimize HPV vaccination in young people, especially males, communication strategies are needed to motivate adolescents to get themselves vaccinated. Texting has been demonstrated to be a feasible, popular, and effective method of sexual health promotion to young people with a relatively low withdrawal rate, positive feedback, and an observed improvement in sexual health knowledge and STI testing (12). Social media communication strategies are a new and potentially effective channel for communicating public health messages about HPV vaccine that are also likely to increase HPV initiation and completion among adolescent girls in addition to boys.

According to the NC Immunization Registry, as of March 8, 2011, only 2% of boys ages 9-13 had received at least one dose of HPV vaccine. In the investigators continuity clinic less than 50 percent of adolescents are fully immunized. This project will identify social behavioral, emotional, and cognitive correlates and predictors that help explain why teens pursue, complete, and do not complete HPV vaccination, and develop a social media communication intervention collaboratively with teens to increase HPV vaccine initiation and completion.

ELIGIBILITY:
Inclusion Criteria:

* incomplete immunization

Exclusion Criteria:

* complete immunization

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescent males and females age 11-21 at a Pediatric clinic
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2015-11-09 (Actual); Study Completion 2016-07-05 (Actual)

PRIMARY OUTCOMES:
HPV vaccination uptake | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Coyne-Beasley, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Pediatric Clinic, Chapel Hill, North Carolina, United States